CLINICAL TRIAL: NCT02139618
Title: A Double-blind Randomized-controlled Trial to Assess the Efficacy of Methyl Aminolevulinate + Daylight vs Placebo + Daylight in Patients With Facial Photodamage
Brief Title: Efficacy of Methyl Aminolevulinate + Daylight in Patients With Facial Photodamage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación Dermabase (Other)
Collaborators: Grupo de Investigacion Dermatologica (GRID) (Unknown); IPS Universitaria-Universidad de Antioquia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-01INT
Record Dates: First submitted 2014-04-29; First posted 2014-05-15 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Facial Photodamage
Keywords: Randomized-controlled-trial; Methyl-Aminolevulinate; Daylight; Photodynamic-therapy
MeSH Terms: interventions — methyl 5-aminolevulinate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methyl Aminolevulinate (MAL) (Experimental): 1 gram of Topical Methyl Aminolevulinate (MAL) applied to the whole face 30 minutes before sun exposure for 2 hours (3 sessions , 2 to 4 weeks apart)
  Interventions: Drug: Methyl Aminolevulinate (MAL)
- Placebo (Placebo Comparator): 1 gram of placebo cream applied to the whole face 30 minutes before sun exposure for 2 hours (3 sessions , 2 to 4 weeks apart)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methyl Aminolevulinate (MAL)
  Other Names: Metvix®
  Arms: Methyl Aminolevulinate (MAL)
Drug: Placebo
  Other Names: Vehicle
  Arms: Placebo

SUMMARY:
Treatment of actinic damage has included multiple procedures but to date there is limited scientific evidence to support the preferential use of one of these therapies according to their efficacy, safety and pain tolerance by patients. This study aims to assess the efficacy of methyl aminolevulinate + daylight vs placebo + daylight to treat facial photodamage

ELIGIBILITY:
Inclusion Criteria:

* Adults with symmetric facial photodamage grade 2 or 3 (Dover´s scale)
* Patients willing to participate
* Signed informed consent

Exclusion Criteria:

* Pregnant or nursing females
* Subjects with any photosensitizing disorder
* Any active infectious skin disorder
* History of herpes simplex in the face
* Subjects with less than 6 months of any previous rejuvenation interfering treatments
* History of systemic isotretinoin in the last year
* Subjects requiring concurrent treatment that would interfere with study objectives and/or assessments
* History of hypersensitivity reactions
* Activities with high sun exposure during 48 hours after treatment
* Clinical suspicion of any systemic or local malignancy

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Global photodamage improvement | 1 month after third session
  The primary outcome is global photodamage improvement 1 month after the third daylight PDT session, according to Dover´s photodamage scale.

SECONDARY OUTCOMES:
Pain measurement | After 2 hours of sun exposure in each session
  Pain evaluation with the visual analogue scale after 2 hours of sun exposure in each of the sessions performed (Sessions 1, 2 and 3).
Specific Photodamage score | 1 month after the third session
  Specific photodamage severity score for fine lines, coarse lines, tactile roughness, mottled pigmentation, sallowness, and erythema one month after the third daylight PDT session, according to Dover´s photodamage scale.
Sun irradiance and illuminance quantification | During the 2 hours of each session
  Sun irradiation and illuminance quantification during exposure
Adverse events | From recruitment until 1 month after the third session
  Any adverse event
Therapy tolerance | 1 week after sessions 1,2 and 3
  Therapy tolerance will be recorded with a scale that includes a 4-grade severity score for oozing, erythema, oedema, desquamation, pigmentation, and vesiculation.
Quality of life assessment (Skindex-29 Instrument) | Basal and 1 month after the third session
  Quality of life assessment (Skindex-29 Instrument)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Sanclemente, Dr, Principal Investigator — Universidad de Antioquia. Medellin, Colombia
Locations (1):
- IPS Universitaria, Medellín, Antioquia, Colombia